CLINICAL TRIAL: NCT05179278
Title: Impact of a PROgram of Cardiovascular Nurse interventionS in a VALVular haEmodynamic Unit (PROCESS-VALVE) on Quality Indicators: a Quasi-experimental Ambispective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIBSP-CEH-2020-140
Record Dates: First submitted 2021-08-05; First posted 2022-01-05 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2023-05

CONDITIONS: Valvular Heart Disease
Keywords: valvular heart disease; nurse consultation; health indicators; post-surgical follow-up
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: post-surgical face-to-face follow up consultation (Experimental)
  Interventions: Other: Post-surgical nurse follow-up
- Control Group: post-surgical telephone follow up consultation (Experimental)
  Interventions: Other: Post-surgical nurse follow-up

INTERVENTIONS:
Other: Post-surgical nurse follow-up — Follow-up face-to-face consultation or follow-up telephone consultation a month after the intervention and telephone consultation at one year

SUMMARY:
The objective of this study is to evaluate the impact of a program of presurgical and postsurgical nurse interventions (PROCESS-VALVE) on quality indicators of the health of patients undergoing percutaneous valve procedures. (waiting times, patient satisfaction, admission times, hospital readmission, mortality, intrahospital complications and nosocomial infections). Design of the study is an ambispective quasi-experimental study. For the control group, data will be collected retrospectively from patients undergoing percutaneous valve procedures who did not receive pre- or postsurgical consultations. The intervention group will comprise those patients who agree to participate in the study and the haemodynamic nurse valve consultation program (PROCESS-VALVE). In addition, the investigators will assess whether a face-to-face postsurgical consultation improved quality indicators compared to postsurgical telephone consultation; for this, a sub-study will be carried out comparing face-to-face or telephone postsurgical follow-up by means of a randomised controlled clinical trial with simple blinding in the intervention group. Study area will be at the Hemodynamic Unit of the Hospital de la Santa Creu i Sant Pau and the study population are chosen patients for percutaneous valvular intervention who attend the pre-surgical consultation at our center. Dependent variable will be the indicators cited in the study aim and the independent variable will be the pre-surgical and post-surgical consultation. In pre-surgical consultation will be done a patient recruitment and will collect sociodemographic and clinical data. At patient will be done an individualized interview with an Ad-Hoc questionnaire and to collect fragility level of study and level of planned connections. In the subsequent follow-up, all pacients will receive a follow-up visit and collect satisfaction and quality indicators. But this pacients will be randomized to telephone follow-up or face-to-face follow up. Sample size has been calculated in 194 to be distributed equally in both groups and the clinical trials groups will be formed by 94 patients in each group The protocol has been modified to an ambispective quasi-experimental study with a subsequent randomization for the type of follow-up (telephone vs face-to-face) due to organizational changes in the participant center.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepted for Heart-Team for percutaneous treatment aortic stenosis/insufficiency and mitral or tricuspid regurgitation
* Patients visited in the pre-surgical nursing consultation

Exclusion Criteria:

* Patients with language barrier
* Patients undergoing emergency surgery for percutaneous treatment aortic stenosis/insufficiency and mitral or tricuspid regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Waiting time | Pre-intervention
  Time since Heart-team accepted until the intervention
Satisfaction assessed by SUCMA 14 Questionnaire | One mounth after intervention
  Use of an adaptation Sucma 14 Questionnaire (in english Questionnaire Satisfaction of Users of Major Ambulatory Surgery). This scale is former for 14 independent questions with 5 options response (likert scale)
Satisfaction assessed by SUCMA 14 Questionnaire | One year after intervention
  Use of an adaptation Sucma 14 Questionnaire (in english Questionnaire Satisfaction of Users of Major Ambulatory Surgery). This scale is former for 14 independent questions with 5 options response (likert scale)
Admission time | During hospital admission ( until the last day of admission)
  Time since intervention until hospital discharge
Rate of Hospital readmission | One mounth after intervention
  Hospital readminission after the intervention for cardiac reasons
Rate of Hospital readmission | One year after intervention
  Hospital readminission after the intervention for cardiac reasons
Rate of Mortality | Into admission time
  Mortality for all reasons (cardiac or other reason)
Rate of Mortality | One mounth after intervention
  Mortality for all reasons (cardiac or other reason)
Rate of Mortality | One year after intervention
  Mortality for all reasons (cardiac or other reason)
Rate of Intrahospital complications | Into admission time
  Procedure complications (vascular, stroke and cardiac complication)
Rate of Intrahospital complications | One mounth after intervention
  Procedure complications (vascular, stroke and cardiac complication)
Rate of Intrahospital complications | One year after intervention
  Procedure complications (vascular, stroke and cardiac complication)
Rate of Nosocomial infection | During hospital admission (until the last day of admission)
  Infection adquired during hospital admission

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valverde Bernal J, Martinez-Soler F, Berga Congost G, Martinez Perez J, Asmarats L, Moreno Arroyo C. Impact of a PROgram of Cardiovascular nursE interventionS in a VALVular haEmodynamic Unit (PROCESS-VALVE) on Quality Indicators: A Quasi-Experimental Ambispective Study. Int J Gen Med. 2023 Sep 20;16:4257-4265. doi: 10.2147/IJGM.S412369. eCollection 2023. PMID 37750105